CLINICAL TRIAL: NCT04390646
Title: Effect of Pulsatile GnRH Therapy on Cognition in Down Syndrome: Randomized Placebo Control Study
Brief Title: GnRH Therapy on Cognition in Down Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nelly Pitteloud (Other)
Responsible Party: Sponsor-Investigator, Nelly Pitteloud, Professor, Head of the Dpt of Endocrinology, Diabetology and Metabolism, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pulse-UP; 700779 (Other: Swissmedic); 2020-00270 (Other: Swissethics)
Record Dates: First submitted 2020-05-05; First posted 2020-05-15 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Down Syndrome; Cognitive Decline; Alzheimer Disease, Early Onset; Olfaction Disorders
Keywords: GnRH
MeSH Terms: conditions — Down Syndrome; Cognitive Dysfunction; Alzheimer Disease; Olfaction Disorders | interventions — Gonadotropin-Releasing Hormone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multicentric randomized double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsatile GnRH pump treatment (Active Comparator)
  Interventions: Drug: GnRH, gonadorelin acetate
- Pulsatile placebo pump treatment (Placebo Comparator)
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: GnRH, gonadorelin acetate — Drug administered by a subcutaneous pump
  Other Names: Lutrelef
  Arms: Pulsatile GnRH pump treatment
Drug: 0.9% NaCl — Drug administered by a subcutaneous pump
  Arms: Pulsatile placebo pump treatment

SUMMARY:
Down syndrome (DS) is the most common chromosomal disorder; with the increasing life expectancy, about 80% of DS adults reach age 65 years old. Early Alzheimer's disease (AD) is the most common cause of death within this population. DS individuals already show AD neuropathology by the age of 30, while it becomes clinically recognized in their late forties. DS subjects also exhibit olfaction defects in adulthood.

To date, there is no treatment available for the cognitive or olfactory defects in DS. The development of an effective treatment targeting cognitive dysfunction in DS adolescents/adults would be warranted.

GnRH, a decapeptide secreted by hypothalamic neurons is the pilot light of reproduction in all mammals. Pulsatile GnRH acts on the gonadotrophs via the GnRH receptor (GNRHR) in the pituitary gland to stimulate LH and FSH, which themselves will act on the gonads to produce gametes and steroids. However, GNRHR are also expressed in cerebral cortex, hippocampus, amygdala, habenula, olfactory structures, and adrenal gland, suggesting that GnRH may have a role beyond reproduction.

Recently, GnRH has been shown to be involved in the process of ageing and lifespan control. Notably, in murine models, GnRH acts as an anti-ageing factor, independent of sex hormones. While ageing is characterized by hypothalamic inflammation and diminished neurogenesis, particularly in the hypothalamus and the hippocampus, GnRH was able to promote adult neurogenesis.

The regulation of GnRH secretion is complex and involves hormonal, neuronal input, and environmental factors.

Prévot et al. recently explored cognition within the Ts65Dn model and showed an age-dependent loss of the ability to recognize new objects. Also, these mice exhibit defects in olfaction. Given the role of GnRH in anti-aging mice model, pulsatile GnRH or continuous GnRH infusion (leading to desensitization of the GNRHR) were given to the Ts65Dn mice for two weeks. Amazingly, pulsatile but not continuous GnRH therapy was able to recover cognitive and olfaction defects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of trisomy 21
* Verbal expression (ability to follow the procedures of the study)
* Consent to a non-hormonal contraception during the whole duration of the study For women: intra-uterine device with copper, a prior tubal ligation or condoms for the partner For men: condoms or vasectomy

Exclusion Criteria:

* Acute illness (clinical or biochemical findings suggesting acute illness/hospitalization)
* Chronic alcohol abuse, illicit drug use, anabolic steroid abuse, psychotropic drugs reported by caregivers
* Taking medication that modifies hormones: spironolactone, ketoconazole, anticoagulants, corticosteroids, ACTH hormone, psychotropics, including antidepressants, antipsychotics and anticonvulsants.
* Known pituitary adenoma and other hormone-dependent tumours
* Participation in another clinical study
* Intention to become a parent during the course of the study
* Females: ovarian cysts, non-hypothalamic anovulation (i.e. polycystic ovary syndrome), pregnancy or lactation
* Males: hematocrit > 54%
* Contraindications for MRI (e.g. pacemaker, metal clips,etc)
* Participant or his/her legal representative do not want to be informed in case of incidental findings

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cognition | Baseline to end of treatment (Week 24)
  Montreal Cognitive Assessment (MoCA) total score ranges between 0 and 30 (cut-off set at 26 for the healthy population)
  Higher scores reflect better performance.

SECONDARY OUTCOMES:
Dimensional change card sorting task (DCCS) | baseline to end of treatment (Week 24)
  change in score of DCCS to assess executive functions
Paired Associated Learning (PAL, part of the CANTAB battery) | baseline to end of treatment (Week 24)
  change in score of PAL to assess learning
Token test | baseline to end of treatment (Week 24)
  change in score of Token test to assess verbal comprehension
Corsi block tapping task | baseline to end of treatment (Week 24)
  change in score to assess visuospatial memory
Litmus non-word-repetition test | baseline to end of treatment (Week 24)
  change in score of Litmus test to assess phonological abilities
Health-related quality of life SF-12 | baseline to end of treatment (Week 24)
  The health-related quality of life (HRQoL) can be used to measure the effects of healthcare interventions and provide quality-improvement outcomes. The Short Form-12 (SF-12) Health Survey is widely used in measuring HRQoL. SF-12 is a reliable, valid measure in a variety of population groups; it is an equivalent substitute for the SF-36v2 for the summary scales.
  The response to each of the 12 items is weighted separately by the physical and mental component summary (PCS and MCS) regression coefficients and then calculated to give the SF-12 PCS and MCS scores.
Adaptive behavior (Vineland II) - caregiver questionnaire | baseline to end of treatment (Week 24)
  change in score of Vineland II (normed assessment tool that assesses adaptive behavior across the areas of communication, activities of daily living, and socialization).
Glycemia | baseline to end of treatment (Week 24)
  Glucose concentration (mmol/L) is a metabolic parameter.
Insulinemia | baseline to end of treatment (Week 24)
  Insulin concentration (nmol/L) is a metabolic parameter.
Total cholesterol | baseline to end of treatment (Week 24)
  Total cholesterol (mmol/L) is a metabolic parameter.
High density lipoprotein (HDL)-cholesterol | baseline to end of treatment (Week 24)
  HDL-cholesterol (mmol/L) is a metabolic parameter.
Low density lipoprotein (LDL)-cholesterol | baseline to end of treatment (Week 24)
  LDL-cholesterol (mmol/L) is a metabolic parameter.
Triglycerides | baseline to end of treatment (Week 24)
  Triglycerides (mmol/L) is a metabolic parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Pitteloud, MD, Principal Investigator — Endocrinology, Metabolism, Diabetology (CHUV)
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Manfredi-Lozano M, Leysen V, Adamo M, Paiva I, Rovera R, Pignat JM, Timzoura FE, Candlish M, Eddarkaoui S, Malone SA, Silva MSB, Trova S, Imbernon M, Decoster L, Cotellessa L, Tena-Sempere M, Claret M, Paoloni-Giacobino A, Plassard D, Paccou E, Vionnet N, Acierno J, Maceski AM, Lutti A, Pfrieger F, Rasika S, Santoni F, Boehm U, Ciofi P, Buee L, Haddjeri N, Boutillier AL, Kuhle J, Messina A, Draganski B, Giacobini P, Pitteloud N, Prevot V. GnRH replacement rescues cognition in Down syndrome. Science. 2022 Sep 2;377(6610):eabq4515. doi: 10.1126/science.abq4515. Epub 2022 Sep 2. PMID 36048943
- See also: CHUV - Etude Pulse-UP — https://www.chuv.ch/fr/edm/edm-home/recherche/etude-pulse-up-trisomie-21